CLINICAL TRIAL: NCT07175064
Title: Nursing-Led Livelihood Programs and Women's Health: Advancing Sustainable Development Goals on Poverty, Good Health and Well-Being, and Decent Work Among Indigenous Aeta in the Philippines
Brief Title: Nursing-Led Livelihood Programs and Women's Health
Acronym: MMS
Status: Completed | Type: Observational
Sponsor: Angeles University Foundation (Other)
Responsible Party: Principal Investigator, Rudena A. Madayag, Assistant Professor, Angeles University Foundation
Other Study IDs: 2024-CON-Faculty-006
Record Dates: First submitted 2025-09-07; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Nutrition Disorders; Stress, Psychological; Mental Health Issue
Keywords: Community Health Nursing; Women's Health; Indigenous Peoples; Philippines; Empowerment
MeSH Terms: conditions — Nutrition Disorders; Stress, Psychological; Empowerment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Livelihood Program Participants: Adult Aeta women, aged 18 years and older, residing in Sitio Monicayo, Pampanga, who have been active participants in nursing-initiated livelihood programs for at least six months prior to enrollment. Participants were selected based on their involvement in bracelet making, rag making, or liquid dishwashing initiatives facilitated by nursing faculty in partnership with local community leaders.
  Interventions: Behavioral: Nursing-Led Livelihood Programs

INTERVENTIONS:
Behavioral: Nursing-Led Livelihood Programs — A set of community-based livelihood initiatives introduced in 2016 and facilitated by nursing faculty in partnership with local leaders. Activities included bracelet making, rag making, and liquid dishwashing. The programs aimed to provide sustainable income, build women's confidence and skills, and indirectly improve health outcomes by addressing poverty-related social determinants of health.

SUMMARY:
This study aims to evaluate the socioeconomic and health impacts of nursing-led livelihood programs among indigenous women in Sitio Monicayo, Pampanga, Philippines. The programs, initiated in 2016, include bracelet making, rag making, and liquid dishwashing. Using an explanatory sequential mixed methods design, Phase 1 surveys Aeta women to assess changes in household income, employment, and six domains: Program Benefits, Facilitation, Self-Confidence, Resilience, Future Intentions, and Barriers. Nonparametric analyses are used to examine program outcomes. Phase 2 involves semi-structured interviews with a subset of participants to contextualize quantitative results, focusing on nutrition, stress reduction, access to medicines, preventive care, and caregiving. Integration through joint displays is planned to highlight alignment and discordance between survey scores and lived experiences. The study seeks to explore the role of nursing-led livelihood interventions in addressing both economic empowerment and social determinants of health, in alignment with the Sustainable Development Goals on poverty, good health and well-being, and decent work.

DETAILED DESCRIPTION:
This study investigates the socioeconomic and health outcomes of nursing-initiated livelihood programs implemented among indigenous Aeta women in Sitio Monicayo, Pampanga, Philippines. The livelihood programs-bracelet making, rag making, and liquid dishwashing-were introduced in 2016 by nursing faculty in partnership with the local community. The research employs an explanatory sequential mixed methods design.

In Phase 1, a nonrandomized cross-sectional survey is conducted with Aeta women who have participated in the livelihood programs for at least six months. Outcomes include household income change, employment shifts, and six composite domains: Program Benefits, Facilitation, Self-Confidence, Resilience, Future Intentions, and Barriers. Nonparametric analyses (Wilcoxon signed-rank, McNemar-Bowker, Kruskal-Wallis, and Spearman's correlations) are performed using SPSS v29.

In Phase 2, semi-structured interviews are conducted with a purposively selected subgroup of participants to contextualize the quantitative findings. Interviews explore barriers and enablers of participation, and their impact on nutrition, stress reduction, preventive care, and caregiving roles. Thematic analysis follows Braun and Clarke's framework, with member checking used to validate findings. Integration is achieved through joint displays to align, complement, or contrast quantitative and qualitative outcomes.

Data quality assurance: Data entry is checked for completeness and internal consistency. Predefined rules for range and coding consistency are applied across variables. A pilot test is conducted before main data collection to ensure reliability and validity of measures. Source data verification is performed by cross-checking survey and interview records with program participation logs.

Sample size: The sample size (N=25 for survey, n=10 for interviews) is based on available program participants and is designed to capture both breadth and depth of experience.

Statistical analysis plan: The primary quantitative outcomes are household income change and employment shifts. Secondary outcomes include composite scores for empowerment and barriers. Qualitative findings are coded inductively and deductively, and integrated with quantitative data to explain mechanisms and identify discordances.

This study was reviewed and approved by the Angeles University Foundation Ethics Review Committee (2024-CON-Faculty-004).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Member of the Aeta community in Sitio Monicayo, Pampanga, Philippines
* Participation in at least one nursing-initiated livelihood program (bracelet making, rag making, or liquid dishwashing) for a minimum of six months
* Willing and able to provide informed consent

Exclusion Criteria:

* Not a resident of Sitio Monicayo or not part of the Aeta community
* Did not participate in the livelihood programs or participated for less than six months
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as female are eligible to participate.
Study Population: Participants were indigenous Aeta women residing in Sitio Monicayo, Pampanga, Philippines, who engaged in nursing-initiated livelihood programs introduced in the community in 2016. The programs were facilitated by nursing faculty in collaboration with local leaders as part of a long-term community health partnership.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Household Income Change | (pre-program, recalled) and at enrollment (current, 2024)
  Change in reported monthly household income before and after participation in livelihood programs, measured using self-reported survey data. Analyzed using Wilcoxon signed-rank test.
Employment Status Shift | From pre-program participation (recalled baseline) to current status at enrollment (2024)
  Change in primary employment status (self-employment, wage work, farming/fishing, or unemployed) before and after program participation, measured using categorical survey data. Analyzed using McNemar-Bowker test.

SECONDARY OUTCOMES:
Program Benefits Score | At enrolment (2024)
  Composite score based on a 5-item questionnaire developed for this study, using a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree), Range: 1-5.
  Interpretation: Higher scores indicate greater perceived program benefits (better outcome).
Self-Confidence and Skill Development Score | At enrolment (2024)
  Composite score based on a 6-item questionnaire developed for this study, using a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree).
  Range: 1-5.
  Interpretation: Higher scores indicate greater self-confidence and skill development (better outcome).
Facilitation and Partnerships Score | At enrolment (2024)
  Composite score based on a 4-item questionnaire developed for this study, using a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree).
  Range: 1-5.
  Interpretation: Higher scores indicate stronger program facilitation and organizational support (better outcome).
Basic Needs and Economic Resilience Score | At enrolment (2024)
  Composite score based on a 5-item questionnaire developed for this study, using a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree).
  Range: 1-5.
  Interpretation: Higher scores indicate greater ability to meet household needs and manage financial shocks (better outcome).
Future Intentions Score | At enrolment (2024).
  Composite score based on a 3-item questionnaire developed for this study, using a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree).
  Range: 1-5.
  Interpretation: Higher scores indicate stronger plans for sustaining or expanding program participation and work opportunities (better outcome).
Perceived Barriers Score | At enrolment (2024).
  Composite score based on a 6-item questionnaire developed for this study, using a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree).
  Range: 1-5.
  Interpretation: Higher scores indicate greater perceived barriers (worse outcome).

OTHER OUTCOMES:
Qualitative Themes on Health and Wellness Description: Semi-structured interviews with 10 participants exploring perceived effects of program participation on nutrition, stress reduction, preventive care, and psychosoc | At enrolment (2024).
  Semi-structured interviews with 10 participants exploring perceived effects of program participation on nutrition, stress reduction, preventive care, and psychosocial well-being. Thematic analysis used to identify and interpret themes.

CONTACTS AND LOCATIONS:
Overall Officials: Rudena A Madayag, MAN, Principal Investigator — Angeles University Foundation
Locations (1):
- Angeles University Foundation, Angeles City, Pampanga, Philippines

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to the small sample size and the potential risk of re-identification of indigenous Aeta participants. Only aggregate data used in the results publication will be available. De-identified datasets may be shared upon reasonable request to the principal investigator, subject to institutional and ethical approval.

REFERENCES:
- [Background] Braun V, Clarke V. Thematic analysis: A practical guide. London: Sage Publications; 2022.
- [Background] Baker P, Smith JP, Garde A, Grummer-Strawn LM, Wood B, Sen G, Hastings G, Perez-Escamilla R, Ling CY, Rollins N, McCoy D; 2023 Lancet Breastfeeding Series Group. The political economy of infant and young child feeding: confronting corporate power, overcoming structural barriers, and accelerating progress. Lancet. 2023 Feb 11;401(10375):503-524. doi: 10.1016/S0140-6736(22)01933-X. Epub 2023 Feb 7. PMID 36764315
- [Background] Guliman EA, Uy JH. Financial decision-making and women's empowerment: Evidence from rural livelihood programs in the Philippines. Asian Women. 2021;37(3):67-88. doi:10.14431/aw.2021.09.37.3.67.